CLINICAL TRIAL: NCT02362152
Title: The Real Life Topical Field Treatment of Actinic Keratosis Study. An Observational Study Focusing on Patient Reported Outcomes
Brief Title: The Real Life Topical Field Treatment of Actinic Keratosis Study
Acronym: RAPID-ACT
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PICATO-1116
Record Dates: First submitted 2015-02-07; First posted 2015-02-12 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic keratosis; Solar keratosis; Field treatment; Ingenol mebutate; Picato
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Fluorouracil; Imiquimod; Diclofenac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Ingenol mebutate: Adults with actinic keratosis eligible to receive topical treatment with one of the four treatments
  Interventions: Drug: Ingenol mebutate
- 5-fluorouracil: Adults with actinic keratosis eligible to receive topical treatment with one of the four treatments
  Interventions: Drug: 5-fluorouracil
- Imiquimod: Adults with actinic keratosis eligible to receive topical treatment with one of the four treatments
  Interventions: Drug: Imiquimod
- Diclofenac: Adults with actinic keratosis eligible to receive topical treatment with one of the four treatments
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Ingenol mebutate — Topical field treatment as prescribed by dermatologist
  Other Names: Picato
  Groups: Ingenol mebutate
Drug: 5-fluorouracil — Topical field treatment as prescribed by dermatologist
  Other Names: 5-FU
  Groups: 5-fluorouracil
Drug: Imiquimod — Topical field treatment as prescribed by dermatologist
  Groups: Imiquimod
Drug: Diclofenac — Topical field treatment as prescribed by dermatologist
  Groups: Diclofenac

SUMMARY:
This non-interventional, multinational study of topical field treatment of actinic keratosis (AK) aims to collect real-life experience with ingenol mebutate as well as one or two other topical field therapies commonly used in the individual country. Physicians will report baseline characteristics, while the main study focus will be on patient reported outcomes 3-4 weeks after treatment completion (treatment satisfaction, adherence, resource utilization and Health Related Quality of Life.

Dermatology centres in Denmark, Norway, Sweden, the Netherlands, the United Kingdom and Canada will participate.

DETAILED DESCRIPTION:
Actinic keratosis (AK) is caused by exposure to UV radiation and has the potential to regress to normal skin or to squamous cell carcinoma. AK treatment options include cryotherapy for solitary lesions and topical field therapy or photodynamic therapy for lesions in an area of sun-damaged skin. This prospective, non-interventional, multinational study aims to describe and compare in a real-life setting the treatment satisfaction, treatment adherence, resource utilization and quality of life during topical field treatment of AK with 5-fluorouracil, imiquimod, diclofenac and ingenol mebutate.

Dermatology centres in Denmark, Sweden, Norway, Canada, the United Kingdom and the Netherlands will aim to include a total of approximately 1600 patients, of which around 100 in each country will be patients scheduled to receive treatment with ingenol mebutate. In each country patients will in addition be recruited for one or two of the other treatment arms, as appropriate in the country.

Only adult patients scheduled to start treatment with imiquimod, 5-fluorouracil, diclofenac or ingenol mebutate who have given informed consent to use data from their medical records for the study and to report study data themselves will be included and followed for the duration of the scheduled treatment + 3-4 weeks.

Physician will report patient demographics and AK characteristics at baseline. Patients will at baseline report AK Quality of Life, including general attitude regarding sun damaged skin at baseline, and, if applicable, treatment satisfaction and adherence with latest previous AK treatment. At 3-4 weeks after end of treatment, the patients will report treatment satisfaction, adherence, resource utilization, health related Quality of Life.

Treating physicians report drug-related Adverse Events in accordance with national laws and regulations and normal clinical practice.

ELIGIBILITY:
Inclusion Criteria: Patients eligible to receive topical treatment with one of the following for treatment of actinic keratosis at the discretion of the dermatologist: Ingenol mebutate, 5-fluorouracil, imiquimod, diclofenac. Informed consent.

-

Exclusion Criteria: Any on-going treatments at study start with ingenol mebutate, 5-fluorouracil, imiquimod or diclofenac; other topical treatment for AK in treatment area; pregnancy or planned pregnancy within treatment period.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with actinic keratosis planned to receive treatment with ingenol mebutate, 5-fluorouracil, imiquimod or diclofenac at the discretion of the dermatologist (and patient).
Sampling Method: Non-Probability Sample
Enrollment: 1168 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction | 3-4 weeks after end of treatment
  Treatment Satisfaction Questionnaire of Medication TSQM 9

SECONDARY OUTCOMES:
Adherence | 3-4 weeks after end of treatment
  Morisky Medication Adherence Scale
Health Related Quality of Life EQ-5D-5L | Baseline and 3-4 weeks after end of treatment
  General measure of health outcome
DLQI | Baseline and 3-4 weeks after end of treatment
  Dermatology Life Quality Index
WPAI | 3-4 weeks after end of treatment
  Work Productivity and Activity Impairment Questionnaire
Local Skin Response | Up to 3-4 weeks after end of treatment
  Occurrence and duration of redness of skin, dry skin, burning, or stinging

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Study Director, Study Director — LEO Pharma
Locations (1):
- Lievensberg Ziekenhuis, Bergen op Zoom, Netherlands

IPD SHARING:
Plan to Share IPD: No